CLINICAL TRIAL: NCT06938373
Title: Development and Application of Accurate Detection Technology Based on Multimodal Data of Breast Cancer Comobid Depression
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: MAD-BCD001
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — peripheral venous blood, fecal sample, saliva and residual biopsy tissue or surgical specimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neoadjuvant therapy breast cancer patient cohort
- HR-positive breast cancer cohort under adjuvant treatment
- Advanced triple-negative immunotherapy and HR-positive endocrine therapy cohorts

SUMMARY:
This study is a prospective, observational clinical research aimed at establishing a multimodal database encompassing clinical information and gut microbiome data from a sample of over 1,000 breast cancer patients comorbid with depression. The research involves collecting cohort sample information from breast cancer patients with comorbid depression, as well as fecal, blood, and saliva specimens for metagenomic sequencing, untargeted metabolite detection, and cortisol level analysis, respectively. Based on the collected multimodal data, diagnostic, efficacy prediction, and prognostic survival prediction models for breast cancer with comorbid depression will be developed. Additionally, a precision prediction cloud platform will be designed and deployed to support data upload, model prediction, and result visualization.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed primary breast cancer; Aged 18-80 years; No prior history of malignancy other than breast cancer; Awareness of their breast cancer diagnosis; Karnofsky Performance Status (KPS) score >70; Willing to provide blood, fecal, and saliva samples with signed informed consent.

Exclusion Criteria:

* Physician-diagnosed mental disorders before or after breast cancer diagnosis; Severe chronic somatic diseases (e.g., central nervous system disorders, severe head trauma, substance abuse/dependence, intellectual disability, diabetes, gynecological diseases, cardiovascular diseases, thyroid disorders, etc.); Presence of two or more primary malignancies of different tissue origins; Central nervous system (CNS) metastasis of breast cancer; Clinically diagnosed digestive system diseases (e.g., enteritis, gastritis); Use of antidepressant or anxiolytic therapy during the study; Use of medications that alter gut function or metabolism during the study; Pregnant or lactating women; Radiotherapy or chemotherapy within the past 21 days; Use of antibiotics, probiotics, prebiotics, or synbiotics within 3 months prior to the study; Other reasons deemed unsuitable for participation by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate，ORR | 2025-03-11 to 2027-03-01
  The propotion defined as subjects with complete remission (CR) and partial remission (PR) among all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China